CLINICAL TRIAL: NCT05087030
Title: A Randomised, Double Blind, Multicentre Phase III Study to Assess the Efficacy and Safety of RGB-14-P Compared to Prolia® in Women With Postmenopausal Osteoporosis
Brief Title: Comparative Efficacy and Safety Study of RGB-14-P and Prolia® in Women With Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGB 14 101; 2020 006017 38 (EudraCT Number)
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Biosimilars; Prolia®
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: A double-blind design will be used during the main and transition periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- RGB-14-P (Main period) (Experimental): Randomized participants will receive subcutaneous (SC) injection of RGB-14-P, on Day 1 of Treatment periods 1 and 2.
  Interventions: Drug: RGB-14-P
- Prolia® (Main period) (Active Comparator): Randomized participants will receive SC injection of Prolia®, on Day 1 of Treatment periods 1 and 2.
  Interventions: Drug: Prolia®
- RGB-14-P (Transition period) (Experimental): Re-randomized participants will receive SC injection of RGB-14-P, on Day 1 of Treatment period 3.
  Interventions: Drug: RGB-14-P
- Prolia® (Transition period) (Active Comparator): Re-randomized participants will receive SC injection of Prolia®, on Day 1 of Treatment period 3.
  Interventions: Drug: Prolia®
- RGB-14-P (Continued till transition period) (Experimental): Randomized participants will continue to receive SC injection of RGB-14-P from the main period till Day 1 of Treatment period 3.
  Interventions: Drug: RGB-14-P

INTERVENTIONS:
Drug: RGB-14-P — Participants will receive RGB-14-P into the thigh, abdomen, or upper arm as per the arm assigned.
  Arms: RGB-14-P (Continued till transition period); RGB-14-P (Main period); RGB-14-P (Transition period)
Drug: Prolia® — Participants will receive Prolia® into the thigh, abdomen, or upper arm as per the arm assigned.
  Arms: Prolia® (Main period); Prolia® (Transition period)

SUMMARY:
This study will be conducted to assess the efficacy, pharmacodynamic (PD), safety, tolerability, and immunogenicity of RGB -14- P compared to US-licensed Prolia® in participants with postmenopausal osteoporosis, in a comparative manner.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicentre, multiple fixed-dose, 2-arm parallel-group study that includes 2 periods as:

1. Main period (52 weeks), consists of Treatment Period 1 (26 weeks) and Treatment Period 2 (26 weeks). On Day 1 of Treatment Period 1, prior to dosing, participants will be randomized in a 1:1 ratio to receive either RGB-14-P or Prolia®.
2. Transition Period: consists of Treatment Period 3 (26 weeks). On Day 1 of Treatment Period 3 (Week 52), a subset of participants who received Prolia® during the Main Period will be re-randomized 1:1 to receive either a dose RGB-14-P or Prolia® in a double-blinded manner. A subset of participants continuing in the Transition Period who received RGB-14-P during the Main Period will continue to receive a dose of RGB-14- P but will also follow the randomization procedure to maintain blinding.

All participants will receive the study drugs on 2 occasions (Weeks 0 and 26), on Day 1 of Treatment Periods 1 and 2. Participants continuing to the Transition Period will receive the study drugs on a third-occasion (Week 52), Day 1 of Treatment Period 3. One Treatment Period will take 6 months (26 weeks, 183 days).

ELIGIBILITY:
Inclusion Criteria:

* Participant is an ambulatory postmenopausal woman, diagnosed with osteoporosis, able to walk, and not bedridden
* Participant has an absolute BMD consistent with T score ≤ 2.5 and ≥ 4.0 at the lumbar spine as measured by dual-energy X-ray absorptiometry (DXA) during the Screening Period and at least 2 lumbar vertebrae (from L1 to L4) must be evaluable by DXA
* Participant has body weight ≥ 50 and ≤ 90 kg at the Screening Period

Participants must meet the following criteria to be enrolled in the Transition Period:

- Have been enrolled, received both doses of the test drug, and completed the scheduled Main Period (up to Week 52) of the RGB-14-101 study

Exclusion Criteria:

* Participant has a history and/or presence of a severe or more than two moderate vertebral fractures as determined by central reading of lateral spine X-ray during the Screening Period
* Participant has a history and/or presence of hip fracture
* Participant has a history and/or presence of atypical femur fracture
* Participant presents with an active healing fracture
* Participant has a bilateral hip replacement (unilateral is allowed if the other hip is evaluable with DXA)
* Participant has a vitamin D deficiency
* Participant has hypocalcaemia or hypercalcemia at the Screening Period
* Participant has a history and/or presence of bone metastases, renal osteodystrophy, osteomyelitis, any metabolic, endocrine or traumatic bone disease
* Participant has a current uncontrolled status of hypothyroidism or hyperthyroidism
* Participant has a history (within 5 years prior to Screening) and/or current hypoparathyroidism or hyperparathyroidism
* Participant has malignancy within 5 years before Screening
* Participant has a history and/or presence of significant cardiac disease
* Participant has a known intolerance or malabsorption of calcium or vitamin D supplements
* Participant shows contraindications to denosumab therapy (e.g., hypocalcaemia), or calcium or vitamin D supplementation before starting test drug administration
* Participant has a latex allergy
* Participant has a history and/or presence of osteonecrosis of the jaw (ONJ) or risk factors for ONJ such as invasive dental procedures
* Participant has history and/or presence of osteonecrosis of the external auditory canal
* Participant requiring ongoing use of any osteoporosis treatment
* Participant has previously received denosumab or biosimilar denosumab
* Participant has weight or girth measurements which may preclude accurate DXA measurements
* Participant has an active infection, including, but not limited to severe acute respiratory syndrome coronavirus-2, hepatis B, hepatitis C and human immunodeficiency virus infections during the Screening Period

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 473 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (4):
  - Miami Clinical Research, Miami, Florida
  - Global Health Research Center, Miami Lakes, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Excel Clinical Research - Internal Medicine, Las Vegas, Nevada
- Bulgaria (10):
  - Medical Center Hera EOOD - Rheumatology Office, Sofia, Sofia-Grad
  - Medical Center Medconsult Pleven, Pleven
  - UMHAT Kaspela, Plovdiv
  - DKC "Sveti Georgi", Plovdiv
  - UMHAT Kaspela (Endocrinology/metabolic disease), Plovdiv
  - UMHAT Pulmed - Reumathology, Plovdiv
  - UMHAT Plovdiv, Plovdiv
  - Medical Center - Teodora EOOD, Rousse
  - Medical Center Excelsior, Sofia
  - "DCC XVII-Sofia" EOOD, Sofia
- Czechia (7):
  - APAVAR Lekarna, Ostrava, Ostrava-město
  - FN Hradec Kralove, Hradec Králové
  - Klatovska nemocnice, a.s., Klatovy
  - Fakultni nemocnice Plzen, Pilsen
  - Revmatologicky ustav, Prague
  - Affidea Praha s.r.o., Prague
  - Fakultni nemocnice v Motole, Prague
- Hungary (6):
  - BAZM KKH EOK Szt Ferenc Tagkh, Miskolc, Borsod-Abauj Zemplen county
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar
  - Qualiclinic Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Csongrad Megyei Dr Bugyi Istvan Korhaz, Szentes
- Italy (3):
  - IRCCS Policlinico San Matteo, Università degli studi di Pavi, Pavia
  - Azienda Ospedaliera di Perugia - Ospedale Santa Maria della, Perugia
  - Azienda Ospedaliero Universitaria Integrata Verona, Veneto
- Poland (17):
  - Barbara Rewerska Diamond Clin., Krakow, Lesser Poland Voivodeship
  - Zespol Poradni Specjalistycznych REUMED, Filia nr 1 Wallenroda, Lublin, Lublin Voivodeship
  - Lubelskie Centrum Diagnostyczne, Świdnik, Lublin Voivodeship
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw, Masovian Voivodeship
  - Komisja Bioetyczna przy OIL w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Nasz Lekarz Osrodek Badan Klinicznych, Bialystok, Podlaskie Voivodeship
  - ClinicMed Daniluk, Nowak Sp. J, Bialystok, Podlaskie Voivodeship
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Centrum Medyczne Pratia Katowice, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Oswiecimskie Centrum Badan Klinicznych, Oświęcim
  - RCMed Oddzial Sochaczew, Sochaczew
  - RCMed, Sochaczew
  - Medycyna Kliniczna, Warsaw
  - RCMed Oddział Warszawa, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw
- Spain (6):
  - H. Ntra. Sra. de la Esperanza, Santiago de Compostela, A Coruña
  - Corporacio Sanitaria Parc Tauli de Sabadell - Servicio de reumatologia, Sabadell, Barcelona
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Centro Medico Instituto Palacios, Madrid
  - Clinica Gaias Santiago, Santiago de Compostela
- Ukraine (6):
  - Medychnyi tsentr tovarystva z obmezhenoyu vidpovidalnistyu "Medbud-Klinik", Kyiv, Kyïv
  - Derzhavna ustanova "Instytut herontolohii imeni D.F. Chebotarova Natsionalnoi akademii medychnykh nauk Ukrainy, Kyiv, Kyïv
  - Vinnytska oblasna klinichna likarnia im. M.I. Pyrohova, Vinnytsia, Vinnytsia Oblast
  - Naukovo-doslidnyi instytut reabilitatsii osib z invalidnistiu (navchalno-naukovo-likuvalnyi kompleks) Vinnytskoho natsionalnoho medychnoho universytetu im. M.I. Pyrohova, Vinnytsia, Vinnytsia Oblast
  - Kyivska klinichna likarnia na zaliznychnomu transporti #2 filii "Tsentr okhorony zdoroviya" AT "Ukrayinska Zaliznytsia", Kiyiv
  - Med tsentr TOV "Tsentr simeinoi medytsyny plius", Kiyiv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 21-September-2021 (first subject first visit) to 15-November-2023 (last subject last visit).
Pre-assignment Details: A total 473 participants were randomized in this study. The screening period was up to 35 days. ICF was signed prior to screening procedures. Subjects received study drug in a randomized order. All study assessments were performed as per the schedule of assessments.
Groups:
- Main Period: RGB-14-P: Participants received RGB-14-P as subcutaneous (SC) injection on Day 1 of Treatment Period 1 (Week 0) and Treatment Period 2 (Week 26).
- Main Period: Prolia®: Participants received Prolia® as SC injection on Day 1 of Treatment Period 1 (Week 0) and Treatment Period 2 (Week 26).
- Transition Period: RGB-14-P to RGB-14-P: Participants who received RGB-14-P during the main period were re-randomized to receive RGB-14-P as SC injection on Day 1 of Treatment period 3 (Week 52).
- Transition Period: Prolia® to RGB-14-P: Participants who received Prolia® during the main period were re-randomized and received RGB-14-P as SC injection on Day 1 of Treatment period 3 (Week 52).
- Transition Period: Prolia® to Prolia®: Participants who received Prolia® during the main period were re-randomized and received Prolia® as SC injection on Day 1 of Treatment period 3 (Week 52).
Period: Main Period (Week 0 to Week 52)
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Started | 242 | 231 | 0 | 0 | 0
Completed | 225 | 211 | 0 | 0 | 0
Not Completed | 17 | 20 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 13 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Subject's Personal Reason | 0 | 2 | 0 | 0 | 0
Not completed — Exclusion criteria met | 1 | 0 | 0 | 0 | 0
Not completed — Study Objective Confounded By Monoclonal Gammopathy | 1 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 0 | 0
Period: Transition Period (Week 52 to Week 78)
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Started | 0 | 0 | 63 | 62 | 63
Completed | 0 | 0 | 63 | 62 | 62
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised all participants to whom the investigational medicinal product (IMP) has been randomized.
  Main period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Total
Number analyzed (Participants) | 242 | 231 | 473
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (5.20) | 66.8 (4.91) | 66.7 (5.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 231 | 473
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 22 | 40
  Not Hispanic or Latino | 223 | 209 | 432
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 2 | 2
  White | 241 | 229 | 470
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline (%CfB) in Lumbar Spine Bone Mineral Density (BMD)
Description: Percentage change from baseline in lumbar bone BMD was assessed. BMD at the lumbar spine was measured by dual-energy x-ray absorptiometry (DXA). This outcome measure was assessed for main period.
Time Frame: Week 52
Population: The Full analysis set (FAS) included all participants to whom the investigational medicinal product (IMP) has been randomized. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia®
Number analyzed (Participants) | 222 | 206
Percentage change from baseline | 5.68 (3.535) | 5.19 (4.118)
Statistical Analysis 1: Comparison: Main Period: RGB-14-P vs Main Period: Prolia®; Test type: Non-Inferiority — The analysis was performed with an ANCOVA model with %CfB in lumbar spine BMD at Week 52 as the dependent variable, covariates were treatment arm (RGB-14-P and US-licensed Prolia); ANCOVA; Estimated Difference = 0.18, 90% CI 2-sided [-0.465 to 0.826]
Statistical Analysis 2: Comparison: Main Period: RGB-14-P vs Main Period: Prolia®; Test type: Superiority — Non-Superiority Test; ANCOVA; Estimated Difference = 0.55, 90% CI 2-sided [-0.099 to 1.191]

2. Primary Outcome: Area Under the Effective Curve (AUEC) After the First Dose Until Day 183 of %CfB in Serum Type I Collagen C-telopeptide (sCTX)
Description: The AUEC of %CfB in sCTX of RGB-14-P was assessed as part of pharmacodynamics parameter with US-licensed Prolia® in female participants was demonstrated with postmenopausal osteoporosis. This outcome measure was assessed for main period only.
Time Frame: Week 26
Population: The pharmacodynamic analysis set included all participants in the safety population with at least one evaluable pharmacodynamic parameter (%CfB and AUEC) and not had any protocol deviations that have a relevant impact on sCTX or serum Prokollagen Typ 1 N-terminales Propeptid (P1NP) results included in the pharmacodynamic parameter calculation. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL*day
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia®
Number analyzed (Participants) | 208 | 196
mg/dL*day | 14609.67 (3142.086) | 14134.86 (7331.714)
Statistical Analysis 1: Comparison: Main Period: RGB-14-P vs Main Period: Prolia®; Comparison between Study Treatment Groups; Test type: Other; p = 0.494, ANCOVA; Geometric mean ratio = 1.01, 95% CI 2-sided [0.978 to 1.046]

3. Secondary Outcome: %CfB in Total Hip BMD
Description: %CfB in total hip BMD was assessed.
Time Frame: Weeks 26, 52 and 78
Population: The FAS included all participants to whom the IMP has been randomized. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure and 'number analyzed in each row' signifies participants with available data that were analyzed for specific timepoint.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 225 | 211 | 63 | 62 | 63
Percentage change from baseline
  Week 26: number analyzed (Participants) | 225 | 211 | 62 | 58 | 62
  Week 26 | 2.42 (2.659) | 2.69 (2.519) | 2.46 (2.712) | 2.81 (2.607) | 3.35 (2.559)
  Week 52: number analyzed (Participants) | 220 | 205 | 63 | 60 | 63
  Week 52 | 3.42 (2.916) | 3.49 (2.872) | 3.03 (3.103) | 3.36 (2.696) | 4.21 (3.452)
  Week 78: number analyzed (Participants) | 0 | 0 | 62 | 62 | 60
  Week 78 |  |  | 4.24 (3.381) | 4.12 (3.128) | 4.95 (3.849)
Statistical Analysis 1: Comparison: Main Period: RGB-14-P vs Main Period: Prolia®; at Week 26; Test type: Other; p = 0.199, Mixed model repeated measures; Estimated difference = -0.31, 95% CI 2-sided [-0.792 to 0.165]
Statistical Analysis 2: Comparison: Main Period: RGB-14-P vs Main Period: Prolia®; At Week 52; Test type: Other; p = 0.543, mixed model repeated measures; Estimated difference = -0.16, 95% CI 2-sided [-0.680 to 0.358]

4. Secondary Outcome: %CfB in Lumbar Spine BMD
Description: %CfB in lumbar spine BMD was assessed.
Time Frame: Weeks 26 and 78
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 227 | 218 | 63 | 62 | 63
Percentage change from baseline
  Week 26: number analyzed (Participants) | 227 | 218 | 62 | 61 | 63
  Week 26 | 3.56 (3.747) | 3.45 (4.227) | 3.98 (3.185) | 3.39 (3.848) | 3.68 (4.979)
  Week 78: number analyzed (Participants) | 0 | 0 | 63 | 62 | 60
  Week 78 |  |  | 7.03 (3.828) | 7.06 (4.327) | 7.09 (4.240)
Statistical Analysis 1: Comparison: Main Period: RGB-14-P vs Main Period: Prolia®; Week 26; Test type: Other; p = 0.929, mixed model for repeated measures; Estimated Difference = 0.03, 95% CI 2-sided [-0.703 to 0.769]

5. Secondary Outcome: %CfB in Femoral Neck BMD
Description: %CfB in femoral neck BMD was assessed by DXA.
Time Frame: Weeks 26, 52 and 78
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 225 | 211 | 63 | 62 | 63
Percentage change from baseline
  Week 26: number analyzed (Participants) | 225 | 211 | 62 | 58 | 62
  Week 26 | 1.88 (3.040) | 1.94 (3.610) | 1.60 (2.833) | 2.21 (3.296) | 2.35 (4.057)
  Week 52: number analyzed (Participants) | 220 | 205 | 63 | 60 | 63
  Week 52 | 2.42 (3.687) | 2.64 (3.751) | 1.95 (3.621) | 2.60 (3.127) | 3.24 (4.549)
  Week 78: number analyzed (Participants) | 0 | 0 | 63 | 62 | 60
  Week 78 |  |  | 3.08 (4.259) | 3.06 (3.337) | 4.04 (4.764)

6. Secondary Outcome: Number of Participants With Vertebral Fragility Fracture
Description: Number of participants with vertebral fragility fracture was assessed. Information on vertebral fractures was centrally collected through the evaluation of lateral thoraco-lumbar spine X-ray.
Time Frame: Weeks 52 and 78
Population: The FAS included all participants to whom the IMP has been randomized. Here, 'number analyzed in each row' signifies the participants with available data that were analyzed for specific timepoint for that outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 242 | 231 | 63 | 62 | 63
Participants
  Week 52: number analyzed (Participants) | 242 | 231 | 0 | 0 | 0
  Week 52 | 4 | 8 |  |  |
  Week 78: number analyzed (Participants) | 0 | 0 | 63 | 62 | 63
  Week 78 |  |  | 3 | 4 | 2

7. Secondary Outcome: Number of Participants With Non-vertebral Fragility Fracture
Description: Number of participants with non-vertebral fragility fracture was assessed. Information on non-vertebral fractures was centrally collected through the evaluation of lateral thoraco-lumbar spine X-ray.
Time Frame: Weeks 52 and 78
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 242 | 231 | 63 | 62 | 63
Participants
  Week 52: number analyzed (Participants) | 242 | 231 | 0 | 0 | 0
  Week 52 | 4 | 10 |  |  |
  Week 78: number analyzed (Participants) | 0 | 0 | 63 | 62 | 63
  Week 78 |  |  | 2 | 5 | 3

8. Secondary Outcome: %CfB in Serum Procollagen Type 1 N Terminal Propeptide (P1NP)
Description: %CfB in serum P1NP was assessed as part of pharmacodynamics parameter with US-licensed Prolia® in female participants with postmenopausal osteoporosis.
Time Frame: Weeks 4, 26, 52 and 78
Population: PD analysis set included all participants in safety population with at least one evaluable PD parameter (%CfB and AUEC) and not had any protocol deviations that have a relevant impact on sCTX or serum P1NP results included in PD parameter calculation. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure and 'number analyzed in each row' signifies participants with available data that were analyzed for specific timepoint.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 234 | 220 | 60 | 60 | 62
Percentage change from baseline
  Week 4: number analyzed (Participants) | 234 | 220 | 60 | 59 | 62
  Week 4 | 22.10 (14.905) | 20.22 (15.091) | 19.85 (13.939) | 18.45 (15.835) | 17.31 (15.524)
  Week 26: number analyzed (Participants) | 216 | 211 | 57 | 59 | 60
  Week 26 | 65.92 (17.828) | 62.89 (29.294) | 68.42 (11.693) | 63.41 (42.677) | 66.08 (16.098)
  Week 52: number analyzed (Participants) | 204 | 198 | 60 | 60 | 61
  Week 52 | 65.04 (19.131) | 63.82 (21.712) | 64.86 (16.902) | 66.05 (20.428) | 65.89 (17.651)
  Week 78: number analyzed (Participants) | 0 | 0 | 54 | 59 | 58
  Week 78 |  |  | 64.12 (18.845) | 66.91 (16.816) | 63.08 (21.364)

9. Secondary Outcome: %CfB in Serum Type I Collagen C-telopeptide (sCTX)
Description: %CfB in sCTX was assessed as part of pharmacodynamics parameter with US-licensed Prolia® was assessed in female participants with postmenopausal osteoporosis.
Time Frame: Weeks 4, 26, 52 and 78
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 234 | 220 | 60 | 60 | 62
Percentage change from baseline
  Week 4: number analyzed (Participants) | 234 | 220 | 60 | 59 | 62
  Week 4 | 85.87 (9.567) | 85.38 (15.501) | 84.96 (11.206) | 84.71 (23.071) | 88.08 (5.832)
  Week 26: number analyzed (Participants) | 216 | 211 | 57 | 59 | 60
  Week 26 | 69.74 (23.212) | 61.51 (83.764) | 67.29 (23.572) | 53.23 (147.679) | 71.27 (17.483)
  Week 52: number analyzed (Participants) | 204 | 198 | 60 | 60 | 61
  Week 52 | 62.90 (28.995) | 58.26 (63.927) | 60.41 (31.958) | 53.89 (94.853) | 66.79 (24.151)
  Week 78: number analyzed (Participants) | 0 | 0 | 54 | 59 | 59
  Week 78 |  |  | 58.70 (34.117) | 53.32 (42.855) | 57.38 (30.562)

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: The safety and tolerability of RGB-14-P with US-licensed Prolia® in female participants with postmenopausal osteoporosis was assessed.
Time Frame: Main Period: From screening (Weeks -5 to 0) to Week 52; Transition Period: From Week 52 to Week 78
Population: Safety analysis set included all participants who received at least one full or partial dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 242 | 231 | 63 | 62 | 63
Participants
  Any AE | 161 | 158 | 0 | 0 | 0
  Any TEAEs | 158 | 152 | 30 | 25 | 25
  Any TEAEs severe or worse severity | 8 | 9 | 0 | 1 | 0
  Any treatment related TEAE | 36 | 32 | 2 | 5 | 1
  Any treatment related TEAE severe or worse severity | 1 | 0 | 0 | 0 | 0
  Any serious TEAEs | 7 | 16 | 0 | 0 | 0
  Any serious TEAEs severe or worse severity | 5 | 9 | 0 | 0 | 0
  Any non-serious TEAEs | 158 | 149 | 30 | 25 | 25
  Any AEs leading to participant discontinuation | 2 | 3 | 0 | 0 | 0
  Any TEAEs leading to subject discontinuation | 2 | 3 | 0 | 0 | 0
  Any treatment related TEAE leading to participant discontinuation | 1 | 0 | 0 | 0 | 0
  Any TEAEs leading to discontinuation of IMP | 2 | 2 | 0 | 0 | 0
  Any treatment related TEAE leading to discontinuation of IMP | 1 | 0 | 0 | 0 | 0
  Any fracture TEAE | 9 | 18 | 4 | 3 | 1
  Any fracture TEAE severe or worse severity | 2 | 1 | 0 | 0 | 0
  Any serious fracture TEAEs | 1 | 1 | 0 | 0 | 0
  Any serious fracture TEAEs severe or worse severity | 1 | 1 | 0 | 0 | 0
  Deaths | 0 | 1 | 0 | 0 | 0
  Any AE leading to death | 0 | 1 | 0 | 0 | 0
  Any TEAE leading to death | 0 | 1 | 0 | 0 | 0
  Any injection site reactions | 0 | 2 | 0 | 3 | 1
  Any treatment related serious TEAE | 0 | 0 | 0 | 0 | 0
  Any treatment related serious TEAE severe or worse severity | 0 | 0 | 0 | 0 | 0
  Any treatment related fracture TEAE | 0 | 0 | 0 | 0 | 0
  Any treatment related fracture TEAE severe or worse severity | 0 | 0 | 0 | 0 | 0
  Any treatment related serious fracture TEAE | 0 | 0 | 0 | 0 | 0
  Any treatment related serious fracture TEAE severe or worse severity | 0 | 0 | 0 | 0 | 0
  Any treatment related fatal serious TEAEs | 0 | 0 | 0 | 0 | 0
  Any injection site reactions of CTCAE grade ≥ 3 | 0 | 0 | 0 | 0 | 0
  Any injection site reactions severe or worse severity | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs)
Description: Number of participants with positive ADAs was assessed.
Time Frame: Weeks 0, 2, 4, 26, 28, 30, 52, 54, 56 and 78
Population: Immunogenicity analysis set included all participants in the safety population who had the pre-dose immunogenicity result and at least one available post-baseline immunogenicity assessment. Here, 'number analyzed in each row' signifies the participants with available data that were analyzed for specific timepoint for that outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 239 | 228 | 63 | 62 | 62
Participants
  Week 0 | 0 | 1 | 0 | 0 | 0
  Week 2: number analyzed (Participants) | 236 | 224 | 63 | 60 | 61
  Week 2 | 2 | 0 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 237 | 226 | 63 | 60 | 62
  Week 4 | 0 | 0 | 0 | 0 | 0
  Week 26: number analyzed (Participants) | 227 | 219 | 63 | 62 | 62
  Week 26 | 0 | 0 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 218 | 206 | 60 | 58 | 59
  Week 28 | 0 | 1 | 0 | 0 | 1
  Week 30: number analyzed (Participants) | 220 | 215 | 63 | 62 | 62
  Week 30 | 0 | 1 | 0 | 0 | 1
  Week 52: number analyzed (Participants) | 225 | 208 | 63 | 62 | 61
  Week 52 | 0 | 0 | 0 | 0 | 0
  Week 54: number analyzed (Participants) | 0 | 0 | 62 | 61 | 62
  Week 54 |  |  | 0 | 0 | 1
  Week 56: number analyzed (Participants) | 0 | 0 | 63 | 62 | 61
  Week 56 |  |  | 0 | 0 | 1
  Week 78: number analyzed (Participants) | 0 | 0 | 63 | 62 | 61
  Week 78 |  |  | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Neutralizing Antibodies
Description: Number of participants with positive neutralizing antibodies was assessed.
Time Frame: Weeks 0, 2, 4, 26, 28, 30, 52, 54, 56 and 78
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 2 | 2 | 0 | 0 | 1
Participants
  Week 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 0 |  | 0 |  |  |
  Week 2: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 2 | 1 |  |  |  |
  Week 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Week 26: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1
  Week 28 |  | 1 |  |  | 1
  Week 30: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1
  Week 30 |  | 0 |  |  | 0
  Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Week 54: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Week 54 |  |  |  |  | 1
  Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Week 56 |  |  |  |  | 1
  Week 78: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Titre of ADAs
Description: The immunogenicity of RGB -14- P with US-licensed Prolia® in female participants with postmenopausal osteoporosis was assessed.
Time Frame: Weeks 0, 2, 4, 26, 28, 30, 52, 54, 56 and 78
Population: as for outcome 11
Measure: Median (Full Range); unit: Titre
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
Number analyzed (Participants) | 239 | 228 | 63 | 62 | 62
Titre
  Week 0 | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | 302.0 [302 to 302] | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response.
  Week 2: number analyzed (Participants) | 236 | 224 | 63 | 60 | 61
  Week 2 | 761.0 [60 to 1462] | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response.
  Week 4: number analyzed (Participants) | 237 | 226 | 63 | 60 | 62
  Week 4 | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response.
  Week 26: number analyzed (Participants) | 227 | 219 | 63 | 62 | 62
  Week 26 | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response.
  Week 28: number analyzed (Participants) | 218 | 206 | 60 | 58 | 59
  Week 28 | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | 172.0 [172 to 172] | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | 172.0 [172 to 172]
  Week 30: number analyzed (Participants) | 220 | 215 | 63 | 62 | 62
  Week 30 | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | 211.0 [211 to 211] | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | 211.0 [211 to 211]
  Week 52: number analyzed (Participants) | 225 | 208 | 63 | 62 | 61
  Week 52 | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response.
  Week 54: number analyzed (Participants) | 0 | 0 | 62 | 61 | 62
  Week 54 |  |  | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | 224.0 [224 to 224]
  Week 56: number analyzed (Participants) | 0 | 0 | 63 | 62 | 61
  Week 56 |  |  | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | 152.0 [152 to 152]
  Week 78: number analyzed (Participants) | 0 | 0 | 63 | 62 | 61
  Week 78 |  |  | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response. | NA [NA to NA] — Here, "NA" indicates that titre was not evaluable due to no positive ADA response.

ADVERSE EVENTS:
Time Frame: Main Period: From screening (Weeks -5 to 0) to Week 52; Transition Period: From Week 52 to Week 78
Description: Safety analysis set included all participants who received at least one full or partial dose of IMP.
Arm/Group | Main Period: RGB-14-P | Main Period: Prolia® | Transition Period: RGB-14-P to RGB-14-P | Transition Period: Prolia® to RGB-14-P | Transition Period: Prolia® to Prolia®
All-Cause Mortality (participants affected / at risk) | 0/242 | 1/231 | 0/63 | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 7/242 | 16/231 | 0/63 | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 100/242 | 85/231 | 4/63 | 3/62 | 6/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Period: RGB-14-P (N=242) | Main Period: Prolia® (N=231) | Transition Period: RGB-14-P to RGB-14-P (N=63) | Transition Period: Prolia® to RGB-14-P (N=62) | Transition Period: Prolia® to Prolia® (N=63)
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Endometrial disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Period: RGB-14-P (N=242) | Main Period: Prolia® (N=231) | Transition Period: RGB-14-P to RGB-14-P (N=63) | Transition Period: Prolia® to RGB-14-P (N=62) | Transition Period: Prolia® to Prolia® (N=63)
COVID-19 (Infections and infestations) | 25 (25) | 24 (25) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 23 (29) | 21 (28) | 1 (1) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 23 (34) | 11 (13) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (13) | 11 (17) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 22 (31) | 22 (27) | 3 (3) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (16) | 10 (13) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (9) | 13 (14) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 14 (15) | 4 (5) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT05087030/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT05087030/SAP_001.pdf